CLINICAL TRIAL: NCT04062227
Title: MBDC-The Mindfulness Based Dementia-Care Study
Brief Title: Mindfulness Based Dementia Care Study
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A18-306
Record Dates: First submitted 2019-08-07; First posted 2019-08-20 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2023-10

CONDITIONS: Caregiver Burnout
Keywords: Mindfulness; Dementia
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mindfulness based stress reduction (MBSR) refers to a particular type of attention focused on the present moment, non-judgmental awareness, and acceptance of that experience with openness and curiosity. Mindfulness training was designed to enhance the range and use of coping skills, decrease levels of stress, improve mood, and reduce tendencies to react in maladaptive ways 1-3. Investigators are evaluating a new program, called the Mindfulness Based Dementia-Care (MBDC) in caregivers (CG) for dementia, which combines the traditional approaches with education. The overall objective of this study is to evaluate the program and explore the potential benefits of the Mindfulness Based Dementia-Care (MBDC) program. Investigators are conducting a prospective, pre-post, observational study with members participating in the MBDC program.

ELIGIBILITY:
Inclusion Criteria:

* Must be ages ≥ 18 years
* Must be able to read and understand English
* Participant of the Mindfulness Based Dementia Care (MBDC) Program

Exclusion Criteria:

* There is no exclusion criteria for this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is anyone who is willing and able to attend the MBDC Program.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kashyap, MBBS, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants of the MBDC Program: Mindfulness Based Dementia Care (MBDC) program is an 8 week program for caregivers (CG) of people living with dementia, which combines traditional mindfulness based stress reduction approaches with education.
Period: Overall Study
Arm/Group | Participants of the MBDC Program
Started | 26
Completed | 16
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 26
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 9
  No age information | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Pre-post Scores on the Perceived Stress Scale (PSS)
Description: The Perceived Stress Scale (PSS) scores on a total score. The range of the PSS is 0-40 points. A lower score is indicative of lower stress.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 20
score on a scale | 4.75 (5.74)

2. Secondary Outcome: Change in Pre-post Scores on the Center for Epidemiologic Studies Depression Scale (CES-D)
Description: The CES-D scores on a total score. The range of the CES-D is 0-60 points. A higher score is indicative of the presence of more depression symptoms.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 20
score on a scale | 6.25 (7.14)

3. Other Pre Specified Outcome: Change in Pre-post Scores on the Self-Compassion Scale (SCS)
Description: The SCS scores on a mean score. The range of the SCS is 1-5 points. A higher score is indicative higher self-compassion.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 20
score on a scale | -0.4 (0.42)

4. Other Pre Specified Outcome: Change in Pre-post Scores on the Resilience Scale
Description: The Resilience Scale scores on a total score. The range of The Resilience Scale is 14-98 points. A higher score is indicative of higher resilience.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 20
score on a scale | 0.25 (13.34)

5. Other Pre Specified Outcome: Change in Pre-post Scores on the Zarit Caregiver Burden Scale.
Description: The Zarit Caregiver Burden Scale scores on a total score. The range of the Zarit range is 0-88 points. A higher score is indicative of the presence of a higher level of caregiver burden.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 20
score on a scale | 2.00 (6.50)

6. Other Pre Specified Outcome: Change in Pre-post Scores on the Brief Coping Orientation to Problems Experienced (COPE)
Description: The Brief COPE scores on fourteen subscale scores. Sub-scores are totaled to give a total range [14-112]. Higher scores indicate increased utilization of coping strategy.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 20
score on a scale | -0.60 (1.11)

7. Other Pre Specified Outcome: Change in Pre-follow-up Scores on the Perceived Stress Scale (PSS)
Description: as for outcome 1
Time Frame: baseline, 5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 11
score on a scale | 2.82 (6.79)

8. Other Pre Specified Outcome: Change in Pre-follow-up Scores on the Center for Epidemiologic Studies Depression Scale (CES-D)
Description: as for outcome 2
Time Frame: baseline, 5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 11
score on a scale | 5.91 (7.35)

9. Other Pre Specified Outcome: Change in Pre-follow-up Scores on the Resilience Scale
Description: as for outcome 4
Time Frame: baseline, 5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 11
score on a scale | -4.82 (8.78)

10. Other Pre Specified Outcome: Change in Pre-follow-up Scores on the Zarit Caregiver Burden Scale
Description: as for outcome 5
Time Frame: baseline, 5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 11
score on a scale | 3.00 (3.93)

11. Other Pre Specified Outcome: Change in Pre-follow-up Scores on the Brief Coping Orientation to Problems Experienced (COPE).
Description: as for outcome 6
Time Frame: baseline, 5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants of the MBDC Program
Number analyzed (Participants) | 11
score on a scale | -0.64 (1.30)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Participants of the MBDC Program
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT04062227/Prot_SAP_000.pdf